CLINICAL TRIAL: NCT03813043
Title: Determination Of The 90% Effective Sedation Dose Of Midazolam In Patients Undergoing Diagnostic Upper Gastric-Endoscopy
Brief Title: The 90% Effective Sedation Dose Of Midazolam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Fahad Specialist Hospital Dammam (Other)
Responsible Party: Principal Investigator, Munir Bamadhaj, Anesthesiologist, King Fahad Specialist Hospital Dammam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANS0307
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Gastro-Esophageal Reflux Disease With Ulceration
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Searching the ED90% of Midazolam using Biased coins method in 40 patients undergoing EGD
Masking Description: The result be found out at the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Midazolam (Other): Midazolam 2 mg as started dosage will be used for first patients and for the other patients will receive an predetermined dosage accordingly
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Midazolam injection — Midazolam 2mg iv to be used as starting dose using Biased coins up and down method (BCM)
  Other Names: Dormicum

SUMMARY:
There are no clear conclusive clinical reports defining the adequate effective dose of midazolam in patients undergoing day-case esophageal-gastro-duodenoscopy (EGD). Defining such dosage will facilitate practitioners who are not anesthesia professionals to administer sedative drugs to establish a satisfactory level of moderate sedation. Our first aim is to determine the effective dose for 90% of patients (ED 90) of midazolam undergoing day-case EGD.

DETAILED DESCRIPTION:
Midazolam is widely used in conscious sedation during esophageal-gastro-duodenoscopy (EGD) to increase patient's tolerance and cooperation. Its short duration, cardiorespiratory stability, anxiolytic and amnestic properties makes it the drug of choice for moderate sedation in day case short procedure 1. Therefore, moderate sedation during digestive endoscopy can be administered by endoscopist in safe monitored area while a qualified nurse monitors the level of consciousness and vital sings. The endoscopist's privileges to administer deeper alternative drug, i.e. propofol, might not be provided easily in many centers especially outside the hospital due to certain limitations. However, the patient's and endoscopist's satisfaction might not be achieved easily with the administration of midazolam for moderate sedation. Inappropriate dose will fail to produce amnesia or may cause respiratory side effect and delayed recovery and discharge. Therefore, there are no clear conclusive clinical reports defining the adequate effective dose of midazolam in patients undergoing day case EGD. This is obvious from different dosage used in various studies. In addition, midazolam dosage in adult is rarely based on the body weight during our daily clinical practice. Defining such dosage will facilitate practitioners who are not anesthesia professionals to administer sedative drugs to establish satisfactory level of moderate sedation. Our first aim is to determine the effective dose for 90% of patients (ED 90) of midazolam undergoing day case EGD.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1&2

Exclusion Criteria:

1. Patients with hypersensitivity to midazolam,
2. Age less than 18,
3. Obstructive sleep apnea
4. known or suspected memory impairment,
5. Patients with psychiatric disorders,
6. visual or hearing impairment and pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Defining the ED90% of Midazolam for sedation of EGD | 10 months
  Calculating the effective Midazolam sedative dosage in 90% of patients undergoing EGD

CONTACTS AND LOCATIONS:
Overall Officials: Ahed zeidan, MD, Study Director — King Fahad Specialist Hospital Dammam

IPD SHARING:
Plan to Share IPD: Undecided
Data will be collected inside the electronic system with limited access